CLINICAL TRIAL: NCT04615767
Title: D-chiro-inositol, a Putative Aromatase Inhibitor, Increases Androgen and Reduces Estrogen Levels in Serum of Male Volunteers. A Pilot Study.
Brief Title: D-chiro-inositol Increases Androgens and Reduces Estrogens in Human Serum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AGUNCO Obstetrics and Gynecology Centre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UVittorio1
Record Dates: First submitted 2020-10-29; First posted 2020-11-04 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-01

CONDITIONS: Low Serum Testosterone Levels in Man
Keywords: Testosterone; DHEAS; Estradiol; Estrone; HOMA index; D-chiro-inositol

STUDY DESIGN:
Intervention Model Description: Ten male volunteers are treated daily with 1 g D-chiro-inositol for 30 days (2 capsules containing 500 mg each, twice a day). The serum levels of the detected parameters at the end of treatment are compared to the values found in the volunteers at the baseline, used as controls. Parameters under analysis: Testosterone/Estradiol ratio, Testosterone, dehydroepiandrosterone, estradiol, estrone, glycemia and insulinemia with Homeostatic Model Assessment for Insulin Resistance (HOMA) index, follicle stimulating hormone, luteinizing hormone, D-chiro-inositol and myo-inositol.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- D-chiro-inositol (Experimental): Volunteers are orally administered with 1 g D-chiro-inositol per day (two doses in capsules of 500 mg each, one in the morning and the other one in the evening) for thirty days
  Interventions: Dietary Supplement: D-chiro-inositol

INTERVENTIONS:
Dietary Supplement: D-chiro-inositol — as described previously

SUMMARY:
The aim of this pilot study is to test the effect of a 30 day-D-chiro-inositol oral treatment on a set of clinical parameters (mainly sex hormones) in a group of male volunteers selected by their age and BMI to investigate if D-chiro-inositol acts as an aromatase inhibitor.

DETAILED DESCRIPTION:
This is an open label clinical trial with a dietary supplement carried out in male volunteers selected by their age and BMI. The aim is to test the effect of oral daily treatment with 1 g D-chiro-inositol for 30 days on some clinical parameters, to see if D-chiro-inositol acts as an aromatase inhibitor. Testosterone, estradiol, Testosterone/Estradiol ratio, Dehydroepiandrosterone sulfate, Estrone, glycemia and insulinemia (with calculation of HOMA index), follicle-stimulating hormone, Luteinizing hormone, D-chiro-inositol and Myo-inositol serum concentrations have to be determined before and after D-chiro-inositol administration.

We wish to evaluate if this treatment for one month is able to change the sexual hormone levels, increasing androgens and decreasing estrogens. Furthermore, we wish to control the safety profile of D-chiro-inositol, a well-known molecule, different from the classic aromatase inhibitors. We think that our pilot study can open up new perspectives of research and therapeutic applications for this many-sided molecule.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) range is between 22 and 34 kg/m2, in order to include subjects with normal weight, overweight and obese. Subjects with altered glycemia or hormonal status due to age or weight were enrolled in the study.

Exclusion Criteria:

* Men with poor general health were excluded from the study.

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 10 (Actual)
Dates: Start 2020-10-28 (Actual); Primary Completion 2020-12-06 (Actual); Study Completion 2020-12-16 (Actual)

PRIMARY OUTCOMES:
Improvement of the Testosterone/Estradiol ratio in serum | Thirty days
  Assessment of the D-Chiro-Inositol treatment to increase the Testosterone/Estradiol ratio by detecting these physiological parameters in serum

SECONDARY OUTCOMES:
Dehydroepiandrosterone sulfate | Thirty days
  Detecting the serum levels of Dehydroepiandrosterone sulfate
Estrone | Thirty days
  Detecting the serum levels of Estrone
Homeostatic Model Assessment for Insulin Resistance (HOMA) Index | Thirty days
  Detecting glycemia and insulinemia

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Monastra, Principal Investigator — Systems Biology Group Lab, Rome, Italy
Locations (1):
- Clinica Alma Res, Rome, Italy

REFERENCES:
- [Derived] Monastra G, Vazquez-Levin M, Bezerra Espinola MS, Bilotta G, Lagana AS, Unfer V. D-chiro-inositol, an aromatase down-modulator, increases androgens and reduces estrogens in male volunteers: a pilot study. Basic Clin Androl. 2021 Jun 3;31(1):13. doi: 10.1186/s12610-021-00131-x. PMID 34078260